CLINICAL TRIAL: NCT04381234
Title: Strategies for Asymmetrical Triacetate Dialyzer
Brief Title: Strategies for Asymmetrical Triacetate Dialyzer Heparin-Free Effective Hemodialysis
Acronym: SAFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: NIPRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S61285
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Hemodialysis Complication
Keywords: anticoagulation; clotting; hemodialysis; hemodiafiltration; citrate
MeSH Terms: conditions — Thrombosis | interventions — Kidneys, Artificial; Renal Dialysis; Citric Acid

STUDY DESIGN:
Intervention Model Description: open-label sequential cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATA plus citrate (Experimental): 1.9 m2 ATA membrane (Solacea™-19H, Nipro Corp., Japan) in combination with citrate (1 mM) containing dialysate
  Interventions: Device: dialyzer; Combination Product: hemodialysis with citrate-containing dialysate
- ATA plus predilution hemodiafiltration (Active Comparator): 1.9 m2 ATA membrane (Solacea™-19H, Nipro Corp., Japan), in combination with high volume predilution hemodiafiltration
  Interventions: Device: dialyzer; Other: predilution hemodiafiltration

INTERVENTIONS:
Device: dialyzer — Asymmetric triacetate dialyzer
  Other Names: Solacea™-19H (Nipro Corp., Japan)
Combination Product: hemodialysis with citrate-containing dialysate — acetate-free dialysate
  Other Names: Selectbag citrate (1mM citrate, Baxter)
  Arms: ATA plus citrate
Other: predilution hemodiafiltration — predilution hemodiafiltration
  Arms: ATA plus predilution hemodiafiltration

SUMMARY:
Not all dialysis patients tolerate heparin anticoagulation. Heparin should be avoided in patients at high risk of bleeding. Strategies include saline infusion, citrate-containing dialysate, regional citrate anticoagulation and heparin-coated membranes. We recently studied the combination of a heparin-coated membrane and citrate-containing dialysate, with a success rate of 94% . Although this combination resulted in low rates of clotting, heparin-coated membranes are not ubiquitously available. The quest for easy to perform, safe and affordable heparin-free dialysis is on. Asymmetric cellulose triacetate (ATA) dialyzers have a low degree of platelet contact activation and might be an alternative to heparin-coated dialyzers.

This is a phase II pilot study in maintenance dialysis patients. Study design is a two-arm open-label cross-over study. In Arm 1, patients were dialyzed using a 1.9 m2 ATA membrane (Solacea™-19H, Nipro Corp., Japan) in combination with citrate (1 mM) containing dialysate. In Arm 2, patients were dialyzed with the same 1.9 m2 ATA membrane, in combination with high volume predilution hemodiafiltration. The primary endpoint was the success rate to complete 4 hours of hemodialysis without preterm clotting.

DETAILED DESCRIPTION:
Anticoagulation is one of the supporting pillars of chronic hemodialysis (HD). The optimal anticoagulant regimen provides full anticoagulation of the extracorporeal circuit with minimal systemic effects and comes at an affordable cost. Unfractionated heparin (UFH) has been the standard of care for many years. In several countries, UFH has gradually been replaced by low molecular weight heparins (LMWH). LMWH are easy to use as they can be administered as a bolus injection and reduce membrane fibrin and platelet deposition. Both UFH and LMWH provide adequate anticoagulation of the extracorporeal circuit, at the price of systemic anticoagulation. Apart from bleeding, the administration of unfractionated heparins has also been associated with dyslipidemia, hypoaldosteronism and hyperkalemia, thrombopenia, osteoporosis, pruritus, and hypersensitivity reactions.

Several alternative anticoagulation regimens have been proposed including saline infusion, heparin coating of the dialyzer membrane as well as regional citrate anticoagulation. Regional citrate anticoagulation is performed by infusing citrate into the arterial line of the dialysis tubing to reduce ionized calcium concentrations in order to minimize propagation of the coagulation cascade. Ionized calcium concentrations are restored by calcium supplementation prior to reinfusion of the blood into the patient. The HepZero study suggested that regional citrate anticoagulation is superior to heparin-coated polyacrylonitrile dialyzers (AN69ST; Nephral 300ST, Gambro) and resulted in in significantly greater instantaneous urea nitrogen clearance. While generally safe and adequate, regional citrate anticoagulation requires additional actions during preparatory phase (preparation of citrate and calcium infusion pumps) as well as during the treatment (measurement of ionized calcium).

Recently, acetate-free citrate-containing dialysate concentrates were introduced into clinical practice. Besides the advantages of acetate-free dialysate, this provides a modest local anticoagulant effect inside the dialyzer. Citrate-containing dialysate allowed to reduce heparin dose while maintaining extracorporeal circuit patency and dialyzer clearance. Recently, citrate-containing dialysate and a heparin-coated dialyzer were combined. In one study, non-inferiority to regional citrate anticoagulation was demonstrated

The abovementioned studies demonstrate that hemodialysis without systemic heparinization is feasible. However, such procedures are more cumbersome, require more manpower, additional biochemical testing and/ or more expensive consumables. The aim of the current study is to test two different strategies for systemic heparin-free dialysis with an asymmetrical tri-acetate hemodialyzer.

Trial objectives To evaluate the feasability, safety and adequacy of systemic heparin-free dialysis using an asymmetrical tri-acetate dialyzer membrane, with or without the combination with citrate containing dialysate.

The main objective of the study is to test efficacy of the two study interventions to perform standard duration (i.e. 4 hours) hemodialysis without interruption due to clotting phenomena and without the use of heparin or low molecular weight heparins.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years, or over. No maximum age is defined.
* Providing signed and dated informed consent (ICF)
* Maintenance dialysis (> 3 months of hemodialysis)
* 'Standard' dialysis regimen (three dialysis sessions / week, dialysis duration 4 hours)
* Hemodynamic stability during 4 weeks preceding study period. Hemodynamic instability is defined as any episode of low blood pressure (asymptomatic or symptomatic requiring intervention (bolus fluid infusion, temporarily withholding or reducing ultrafiltration, preterm termination of dialysis session, resuscitation)
* Hemoglobin 9 - 12 g/dl.

Exclusion Criteria:

* Any known medical disorder favoring either bleeding or clotting (e.g. atypical hemolytic uremic syndrome (aHUS), antiphospholipid syndrome, idiopathic thrombocytopenic purpura (ITP), paroxysmal nocturnal hemoglobinuria (PNH))
* Treatment with a vitamin K antagonist
* Treatment with any one of the NOACs (apixaban, rivaroxaban, edoxaban, dabigatran)
* High risk of bleeding according to the criteria of Swartz (12).
* Patients with a known allergic reaction to asymmetric triacetate
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
clinical patency of the hemodialysis extracorporeal circuit | 4 hours
  clotting of the extracorporeal circuit

SECONDARY OUTCOMES:
Clotting of dialyser | 4 hours
  Semi-quantitative clotting score
dialysis adequacy | 4hours
  single pool Kt/V
Reduction ratio uremic retention solutes | 4 hours
  ratio describing the change in serum concentration over the concentration at the beginning of the dialysis session

CONTACTS AND LOCATIONS:
Overall Officials: bjorn D Meijers, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593